CLINICAL TRIAL: NCT03577119
Title: Full-fat Yogurt and Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, Jana Kraft, Principal Investigator, University of Vermont Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 18-0295
Record Dates: First submitted 2018-06-01; First posted 2018-07-05 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Pre-Diabetes
Keywords: Prediabetes; Glucose Tolerance; Bioactive fatty acids; Insulin sensitivity; Diet; Milk fat; Lipid metabolism; Inflammation markers; Fecal microbiota composition; Dairy
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study will employ a controlled, randomized, double-blinded crossover trial comparing two diets.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-fat yogurt (Experimental): Participants will receive a 21-day controlled diet that includes three daily servings of whole (3.25% fat) yogurt (38% of energy from fat, 44% of energy from carbohydrates, and 18% of energy from protein).
  Interventions: Dietary Supplement: Full-fat yogurt
- Non-fat yogurt (Control) (Experimental): Participants will receive a 21-day controlled diet that includes three daily servings of fat-free yogurt (28% of energy from fat, 54% of energy from carbohydrates, and 18% of energy from protein).
  Interventions: Dietary Supplement: Non-fat yogurt

INTERVENTIONS:
Dietary Supplement: Full-fat yogurt — Controlled diet that includes three daily servings of whole (3.25% fat) yogurt.
  Arms: Full-fat yogurt
Dietary Supplement: Non-fat yogurt — Controlled diet that includes three daily servings of fat-free yogurt.
  Arms: Non-fat yogurt (Control)

SUMMARY:
This study determines if substituting full-fat yogurt (i.e., whole, 3.25% fat) for non-fat yogurt in the diet can reduce the risk of type 2 diabetes and inflammation in association with changes in the composition of the gastrointestinal bacteria prediabetic male and female volunteers. The central hypothesis is that dairy fat impacts whole body glucose handling and insulin sensitivity as well as inflammation both directly, and indirectly via influencing the gut microbiota composition.

DETAILED DESCRIPTION:
The overall objective of this study is to determine if substituting full-fat yogurt (i.e., whole, 3.25% fat) for non-fat yogurt in the diet can i) improve whole body glucose handling and insulin sensitivity, ii) modulate systemic inflammation, and iii) induce putatively beneficial changes in the composition of the colonic microbiota in prediabetic men and women. By comparing a diet containing non-fat yogurt with a diet comprising of full-fat yogurt, the investigators will address the following specific hypotheses and aims:

Hypothesis 1: Dietary intake of full-fat yogurt will improve fasting and postprandial markers of glucose homeostasis, insulin sensitivity, and pancreatic cell function. Aim 1: Evaluating the diet-induced changes in blood glucose and endogenous insulin secretion. This will be assessed through a mixed meal tolerance test and oral glucose tolerance test.

Hypothesis 2: Dietary intake of full-fat yogurt will relatively reduce systemic inflammation. Aim 2: Examine diet-induced changes in inflammatory tone. This will be assessed through measurements of circulating (plasma) pro- and anti-inflammatory cytokines, cytokine production assays from in vitro-stimulated peripheral blood mononuclear cells, and plasma stimulated cytokine production in immortalized human cell lines.

Hypothesis 3: A diet containing full-fat yogurt will alter the colonic bacteria structure (e.g. decrease the Firmicutes/Bacteroidetes ratio). Aim 3: Characterize diet-induced alterations in colonic bacteria structure (composition and density) via next-generation sequencing and real-time Polymerase Chain Reaction Assays (PCR).

This study recruits 32 pre-diabetic female and male volunteers (50:50) aged 45-75 using a double-blinded, randomized crossover design to compare two experimental diets, 1) a low-fat diet containing fat-free yogurt (total fat: 28% energy), and 2) a higher fat diet consisting of whole 3.25% fat yogurt (total fat: 38% energy). Fat in the whole yogurt accounts entirely for the arithmetic difference in fat of 10% energy between the two diets. The study will consist of two 21-day experimental diet periods preceded by a 7-day control diet. The total length of study will be 8 weeks. The diet during the control diet periods will be an average U.S. diet to establish a normalized fatty acid intake among the subjects and to standardize the subject's physiologic state before each experimental diet. At the end of the first control period ("run-in") and at the end of each of the experimental diets, a mixed meal tolerance test and an oral glucose test will be performed to assess diet-induced changes in whole-body glucose handling and insulin sensitivity. In addition, blood and stool samples will be collected to examine diet-induced alterations in inflammatory tone and gastrointestinal microflora.

ELIGIBILITY:
Inclusion Criteria:

* Men and women and not expecting major lifestyle changes while on study
* Age 45-75
* Overweight and obesity (BMI 20-45 kg/m2)
* Stable body weight for the last 6 months (no more than a +/- 5% change)
* Diagnosis of prediabetes, defined as either impaired fasting glucose (fasting glucose: 100-125 mg/dL), impaired glucose tolerance (blood glucose levels of between: 140-199 mg/dL 2-hr post 75-g oral glucose tolerance test), and/or a hemoglobin A1C (HbA1C) level ranging from 5.7% to 7.0% (if HbA1C above 6.4%, monotherapy of Metformin)
* Women: Post-Menopausal: no menses previous 12 mos.; Follicular Stimulating Hormone (FSH) > 20 mIU/mL
* Consuming at least 25% of calories from fat (screening will be based an online fat screener:

http://nutritionquest.com/wellness/free-assessment-tools-for-individuals/fat-intake-screener/

* Normal cognition
* Read and understand English
* Have a telephone
* Willing to follow the study coordinator's/manager's and dietitian's instructions

Exclusion Criteria:

* Fasting blood glucose ≥126 mg/dL, HbA1C ≥7.0% without monotheraoy of Metformin
* Subject with any chronic disease, inflammatory disease (e.g., asthma, rheumatoid arthritis, Crohn's disease or inflammatory bowel disease) and previous diagnosis of HIV or hepatitis C
* Pregnant or breastfeeding women or women on hormone replacement therapy (for previous 3 months)
* Intolerance to dairy foods (i.e., lactose intolerance or protein allergy), food allergies, or significant food preferences, dietary restrictions (vegetarian, vegan lifestyle), or food aversions that would interfere with diet adherence
* History of a diagnosed eating disorder
* Known/diagnosed gastrointestinal problems (e.g., inflammatory bowel disease, irritable bowel syndrome, etc.)
* Antibiotics use during the past 6 months
* Habitual use of tobacco or controlled substances, and dietary supplements during the study and 1 month prior to the study
* On medically prescribed diets or following a diet (e.g., to lose weight) or use of obesity or weight-loss treatments such as dietary interventions or pharmacotherapy
* Chronic anti-inflammatory medications, or frequent use (>25% of the time) of over-the-counter medication including laxatives and antacids (subjects with occasional use of allergy or cold medicine, NSAIDS, acetaminophen, or aspirin will be recruited, but these drugs will not be permitted during the study, except for acute administration up to 3 days prior to the outcome variables).
* Waist circumference >40 inches in men and >35 inches in women
* Current diagnosis of uncontrolled hypertension (systolic BP: >160mmHg, diastolic BP: >95mmHg), (may receive treatment for hypertension as long as 1) on a stable regime for the previous 6 wk, and 2) no anticipated change while on the study)
* Untreated hyperlipidemia [may receive treatment for hyperlipidemia (statins) as long as 1) on a stable regime for the previous 6 wk, and 2) no anticipated change while on the study)
* Participation on regular basis in competitive sports or habitual aerobic exercise training, which we will arbitrarily define a consisting of > 3 bouts/wk of aerobic exercise (unable to speak comfortably) for more than 20 min
* Lifestyle or schedule incompatible with the study protocol
* Psychiatric or behavioral conditions that in the view of the principal investigator may present a safety hazard to the participant or interfere with study participation or the ability to follow the intervention protocol

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity and β-cell function: MMTT | Baseline, 4 weeks, and 8 weeks
  Evaluated through mixed meal tolerance test (MMTT) prior to and post experimental diets. Tests will be quantified using the area under the curve (AUC) of the temporal changes in blood glucose, insulin, C-peptide, and incretins (GLP-1 and GIP) using fasting and serial postprandial blood samples. All measurements will be reported as mol/L.
Changes in insulin sensitivity and β-cell function: OGTT | Baseline, 4 weeks, and 8 weeks
  Evaluated through oral glucose tolerance test (OGTT) prior to and post experimental diets. Tests will be quantified using the area under the curve (AUC) of the temporal changes in blood glucose, insulin, C-peptide, and incretins (GLP-1 and GIP) using fasting and serial postprandial blood samples. All measurements will be reported as mol/L.

SECONDARY OUTCOMES:
Changes in inflammatory markers | Baseline, 4 weeks, and 8 weeks
  Evaluated through measurements of circulating (plasma) pro- and anti-inflammatory cytokines, cytokine production assays from in vitro-stimulated peripheral blood mononuclear cells, and plasma stimulated cytokine production in immortalized human cell lines prior to and post experimental diets. Inflammatory markers that will be measured are: interleukins 1beta, 6, 8, and 10 (IL-1beta, IL-6, IL-8, and IL-10), and tumor necrosis factor alpha (TNFalpha). All measurements will be reported as pg/mL.
Changes to Colonic microbiota structure: density | Baseline, 4 weeks, and 8 weeks
  Evaluated through analysis of colonic bacteria structure (composition and density) of specific colonic microbiota prior to and post experimental diets. Density of colonic bacteria will be measured in log copies/ug feces.
Changes to Colonic microbiota structure: relative abundance | Baseline, 4 weeks, and 8 weeks
  Evaluated through analysis of colonic bacteria structure (composition and density) of specific colonic microbiota prior to and post experimental diets. Relative abundance of Taxa of colonic bacteria will be reported as a percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Jana Kraft, PhD, Principal Investigator — University of Vermont
Locations (1):
- Clinical Research Center, University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmberg S, Thelin A. High dairy fat intake related to less central obesity: a male cohort study with 12 years' follow-up. Scand J Prim Health Care. 2013 Jun;31(2):89-94. doi: 10.3109/02813432.2012.757070. Epub 2013 Jan 15. PMID 23320900
- [Background] Kratz M, Baars T, Guyenet S. The relationship between high-fat dairy consumption and obesity, cardiovascular, and metabolic disease. Eur J Nutr. 2013 Feb;52(1):1-24. doi: 10.1007/s00394-012-0418-1. Epub 2012 Jul 19. PMID 22810464
- [Background] Scharf RJ, Demmer RT, DeBoer MD. Longitudinal evaluation of milk type consumed and weight status in preschoolers. Arch Dis Child. 2013 May;98(5):335-40. doi: 10.1136/archdischild-2012-302941. Epub 2013 Mar 18. PMID 23508869
- [Background] Li, S., Field, A., Rimm, E. & Flint, A. Dairy consumption with onset of overweight and obesity among U.S. adolescents. FASEB J 28, 370.7 (2014).
- [Background] Kratz M, Marcovina S, Nelson JE, Yeh MM, Kowdley KV, Callahan HS, Song X, Di C, Utzschneider KM. Dairy fat intake is associated with glucose tolerance, hepatic and systemic insulin sensitivity, and liver fat but not beta-cell function in humans. Am J Clin Nutr. 2014 Jun;99(6):1385-96. doi: 10.3945/ajcn.113.075457. Epub 2014 Apr 16. PMID 24740208
- [Background] Yakoob MY, Shi P, Willett WC, Rexrode KM, Campos H, Orav EJ, Hu FB, Mozaffarian D. Circulating Biomarkers of Dairy Fat and Risk of Incident Diabetes Mellitus Among Men and Women in the United States in Two Large Prospective Cohorts. Circulation. 2016 Apr 26;133(17):1645-54. doi: 10.1161/CIRCULATIONAHA.115.018410. Epub 2016 Mar 22. PMID 27006479
- [Background] Ericson U, Hellstrand S, Brunkwall L, Schulz CA, Sonestedt E, Wallstrom P, Gullberg B, Wirfalt E, Orho-Melander M. Food sources of fat may clarify the inconsistent role of dietary fat intake for incidence of type 2 diabetes. Am J Clin Nutr. 2015 May;101(5):1065-80. doi: 10.3945/ajcn.114.103010. Epub 2015 Apr 1. PMID 25832335
- [Background] Gijsbers L, Ding EL, Malik VS, de Goede J, Geleijnse JM, Soedamah-Muthu SS. Consumption of dairy foods and diabetes incidence: a dose-response meta-analysis of observational studies. Am J Clin Nutr. 2016 Apr;103(4):1111-24. doi: 10.3945/ajcn.115.123216. Epub 2016 Feb 24. PMID 26912494
- [Background] Jensen RG. The composition of bovine milk lipids: January 1995 to December 2000. J Dairy Sci. 2002 Feb;85(2):295-350. doi: 10.3168/jds.S0022-0302(02)74079-4. PMID 11913692
- [Background] Roy CC, Kien CL, Bouthillier L, Levy E. Short-chain fatty acids: ready for prime time? Nutr Clin Pract. 2006 Aug;21(4):351-66. doi: 10.1177/0115426506021004351. PMID 16870803
- [Background] Barber MC, Clegg RA, Travers MT, Vernon RG. Lipid metabolism in the lactating mammary gland. Biochim Biophys Acta. 1997 Aug 16;1347(2-3):101-26. doi: 10.1016/s0005-2760(97)00079-9. No abstract available. PMID 9295156
- [Background] Keeney, M. K., Katz, I. & Allison, M.J. On the probable origin of some milk fat acids in rumen microbial lipids. J Am Oil Chem Soc 39, 198-201 (1962).
- [Background] Jenkins B, West JA, Koulman A. A review of odd-chain fatty acid metabolism and the role of pentadecanoic Acid (c15:0) and heptadecanoic Acid (c17:0) in health and disease. Molecules. 2015 Jan 30;20(2):2425-44. doi: 10.3390/molecules20022425. PMID 25647578
- [Background] Palmquist DL, Lock AL, Shingfield KJ, Bauman DE. Biosynthesis of conjugated linoleic acid in ruminants and humans. Adv Food Nutr Res. 2005;50:179-217. doi: 10.1016/S1043-4526(05)50006-8. No abstract available. PMID 16263431
- [Background] Shingfield KJ, Chilliard Y, Toivonen V, Kairenius P, Givens DI. Trans fatty acids and bioactive lipids in ruminant milk. Adv Exp Med Biol. 2008;606:3-65. doi: 10.1007/978-0-387-74087-4_1. No abstract available. PMID 18183924
- [Background] Bainbridge ML, Cersosimo LM, Wright AD, Kraft J. Content and Composition of Branched-Chain Fatty Acids in Bovine Milk Are Affected by Lactation Stage and Breed of Dairy Cow. PLoS One. 2016 Mar 1;11(3):e0150386. doi: 10.1371/journal.pone.0150386. eCollection 2016. PMID 26930646
- [Background] Calder PC. Dietary modification of inflammation with lipids. Proc Nutr Soc. 2002 Aug;61(3):345-58. doi: 10.1079/pns2002166. PMID 12296294
- [Background] Antoniades C, Bakogiannis C, Tousoulis D, Demosthenous M, Marinou K, Stefanadis C. Platelet activation in atherogenesis associated with low-grade inflammation. Inflamm Allergy Drug Targets. 2010 Dec;9(5):334-45. doi: 10.2174/187152810793938035. PMID 20632958
- [Background] Bohl M, Bjornshave A, Gregersen S, Hermansen K. Whey and Casein Proteins and Medium-Chain Saturated Fatty Acids from Milk Do Not Increase Low-Grade Inflammation in Abdominally Obese Adults. Rev Diabet Stud. 2016 Summer-Fall;13(2-3):148-157. doi: 10.1900/rds.2016.13.148. Epub 2016 Mar 14. PMID 28012280
- [Background] Calder PC, Ahluwalia N, Brouns F, Buetler T, Clement K, Cunningham K, Esposito K, Jonsson LS, Kolb H, Lansink M, Marcos A, Margioris A, Matusheski N, Nordmann H, O'Brien J, Pugliese G, Rizkalla S, Schalkwijk C, Tuomilehto J, Warnberg J, Watzl B, Winklhofer-Roob BM. Dietary factors and low-grade inflammation in relation to overweight and obesity. Br J Nutr. 2011 Dec;106 Suppl 3:S5-78. doi: 10.1017/S0007114511005460. PMID 22133051
- [Background] Cani PD, Osto M, Geurts L, Everard A. Involvement of gut microbiota in the development of low-grade inflammation and type 2 diabetes associated with obesity. Gut Microbes. 2012 Jul-Aug;3(4):279-88. doi: 10.4161/gmic.19625. Epub 2012 May 14. PMID 22572877
- [Background] Lalles JP. Dairy products and the French paradox: Could alkaline phosphatases play a role? Med Hypotheses. 2016 Jul;92:7-11. doi: 10.1016/j.mehy.2016.04.033. Epub 2016 Apr 20. PMID 27241245
- [Background] Misiak B, Leszek J, Kiejna A. Metabolic syndrome, mild cognitive impairment and Alzheimer's disease--the emerging role of systemic low-grade inflammation and adiposity. Brain Res Bull. 2012 Nov 1;89(3-4):144-9. doi: 10.1016/j.brainresbull.2012.08.003. Epub 2012 Aug 18. PMID 22921944
- [Background] Perry VH. Contribution of systemic inflammation to chronic neurodegeneration. Acta Neuropathol. 2010 Sep;120(3):277-86. doi: 10.1007/s00401-010-0722-x. Epub 2010 Jul 20. PMID 20644946
- [Background] Vitale G, Salvioli S, Franceschi C. Oxidative stress and the ageing endocrine system. Nat Rev Endocrinol. 2013 Apr;9(4):228-40. doi: 10.1038/nrendo.2013.29. Epub 2013 Feb 26. PMID 23438835
- [Background] Poynter ME, Daynes RA. Peroxisome proliferator-activated receptor alpha activation modulates cellular redox status, represses nuclear factor-kappaB signaling, and reduces inflammatory cytokine production in aging. J Biol Chem. 1998 Dec 4;273(49):32833-41. doi: 10.1074/jbc.273.49.32833. PMID 9830030
- [Background] Hammond RA, Levine R. The economic impact of obesity in the United States. Diabetes Metab Syndr Obes. 2010 Aug 30;3:285-95. doi: 10.2147/DMSOTT.S7384. PMID 21437097
- [Background] Ferdinand, K. C. et al. Health economics of cardiovascular disease: Defining the research agenda. CVD Prev Control 6, 91-100 (2011).
- [Background] O'Neill S, O'Driscoll L. Metabolic syndrome: a closer look at the growing epidemic and its associated pathologies. Obes Rev. 2015 Jan;16(1):1-12. doi: 10.1111/obr.12229. Epub 2014 Nov 18. PMID 25407540
- [Background] Barbaresko J, Koch M, Schulze MB, Nothlings U. Dietary pattern analysis and biomarkers of low-grade inflammation: a systematic literature review. Nutr Rev. 2013 Aug;71(8):511-27. doi: 10.1111/nure.12035. Epub 2013 Jun 13. PMID 23865797
- [Background] Minihane AM, Vinoy S, Russell WR, Baka A, Roche HM, Tuohy KM, Teeling JL, Blaak EE, Fenech M, Vauzour D, McArdle HJ, Kremer BH, Sterkman L, Vafeiadou K, Benedetti MM, Williams CM, Calder PC. Low-grade inflammation, diet composition and health: current research evidence and its translation. Br J Nutr. 2015 Oct 14;114(7):999-1012. doi: 10.1017/S0007114515002093. Epub 2015 Jul 31. PMID 26228057
- [Background] Panagiotakos DB, Pitsavos CH, Zampelas AD, Chrysohoou CA, Stefanadis CI. Dairy products consumption is associated with decreased levels of inflammatory markers related to cardiovascular disease in apparently healthy adults: the ATTICA study. J Am Coll Nutr. 2010 Aug;29(4):357-64. doi: 10.1080/07315724.2010.10719852. PMID 21041810
- [Background] Labonte ME, Couture P, Richard C, Desroches S, Lamarche B. Impact of dairy products on biomarkers of inflammation: a systematic review of randomized controlled nutritional intervention studies in overweight and obese adults. Am J Clin Nutr. 2013 Apr;97(4):706-17. doi: 10.3945/ajcn.112.052217. Epub 2013 Feb 27. PMID 23446894
- [Background] Bordoni A, Danesi F, Dardevet D, Dupont D, Fernandez AS, Gille D, Nunes Dos Santos C, Pinto P, Re R, Remond D, Shahar DR, Vergeres G. Dairy products and inflammation: A review of the clinical evidence. Crit Rev Food Sci Nutr. 2017 Aug 13;57(12):2497-2525. doi: 10.1080/10408398.2014.967385. PMID 26287637
- [Background] Calder PC. Fatty acids and inflammation: the cutting edge between food and pharma. Eur J Pharmacol. 2011 Sep;668 Suppl 1:S50-8. doi: 10.1016/j.ejphar.2011.05.085. Epub 2011 Jul 28. PMID 21816146
- [Background] Kien CL, Bunn JY, Fukagawa NK, Anathy V, Matthews DE, Crain KI, Ebenstein DB, Tarleton EK, Pratley RE, Poynter ME. Lipidomic evidence that lowering the typical dietary palmitate to oleate ratio in humans decreases the leukocyte production of proinflammatory cytokines and muscle expression of redox-sensitive genes. J Nutr Biochem. 2015 Dec;26(12):1599-606. doi: 10.1016/j.jnutbio.2015.07.014. Epub 2015 Aug 1. PMID 26324406
- [Background] Kien CL, Bunn JY, Poynter ME, Stevens R, Bain J, Ikayeva O, Fukagawa NK, Champagne CM, Crain KI, Koves TR, Muoio DM. A lipidomics analysis of the relationship between dietary fatty acid composition and insulin sensitivity in young adults. Diabetes. 2013 Apr;62(4):1054-63. doi: 10.2337/db12-0363. Epub 2012 Dec 13. PMID 23238293
- [Background] Kien CL, Matthews DE, Poynter ME, Bunn JY, Fukagawa NK, Crain KI, Ebenstein DB, Tarleton EK, Stevens RD, Koves TR, Muoio DM. Increased palmitate intake: higher acylcarnitine concentrations without impaired progression of beta-oxidation. J Lipid Res. 2015 Sep;56(9):1795-807. doi: 10.1194/jlr.M060137. Epub 2015 Jul 8. PMID 26156077
- [Background] Vinolo MA, Rodrigues HG, Nachbar RT, Curi R. Regulation of inflammation by short chain fatty acids. Nutrients. 2011 Oct;3(10):858-76. doi: 10.3390/nu3100858. Epub 2011 Oct 14. PMID 22254083
- [Background] Tan J, McKenzie C, Potamitis M, Thorburn AN, Mackay CR, Macia L. The role of short-chain fatty acids in health and disease. Adv Immunol. 2014;121:91-119. doi: 10.1016/B978-0-12-800100-4.00003-9. PMID 24388214
- [Background] Andoh A, Fujiyama Y, Hata K, Araki Y, Takaya H, Shimada M, Bamba T. Counter-regulatory effect of sodium butyrate on tumour necrosis factor-alpha (TNF-alpha)-induced complement C3 and factor B biosynthesis in human intestinal epithelial cells. Clin Exp Immunol. 1999 Oct;118(1):23-9. doi: 10.1046/j.1365-2249.1999.01038.x. PMID 10540155
- [Background] Sales-Campos H, Souza PR, Peghini BC, da Silva JS, Cardoso CR. An overview of the modulatory effects of oleic acid in health and disease. Mini Rev Med Chem. 2013 Feb;13(2):201-10. PMID 23278117
- [Background] Vassiliou EK, Gonzalez A, Garcia C, Tadros JH, Chakraborty G, Toney JH. Oleic acid and peanut oil high in oleic acid reverse the inhibitory effect of insulin production of the inflammatory cytokine TNF-alpha both in vitro and in vivo systems. Lipids Health Dis. 2009 Jun 26;8:25. doi: 10.1186/1476-511X-8-25. PMID 19558671
- [Background] Carrillo C, Cavia Mdel M, Alonso-Torre S. Role of oleic acid in immune system; mechanism of action; a review. Nutr Hosp. 2012 Jul-Aug;27(4):978-90. doi: 10.3305/nh.2012.27.4.5783. PMID 23165533
- [Background] Jacome-Sosa M, Vacca C, Mangat R, Diane A, Nelson RC, Reaney MJ, Shen J, Curtis JM, Vine DF, Field CJ, Igarashi M, Piomelli D, Banni S, Proctor SD. Vaccenic acid suppresses intestinal inflammation by increasing anandamide and related N-acylethanolamines in the JCR:LA-cp rat. J Lipid Res. 2016 Apr;57(4):638-49. doi: 10.1194/jlr.M066308. Epub 2016 Feb 17. PMID 26891736
- [Background] Jaudszus A, Jahreis G, Schlormann W, Fischer J, Kramer R, Degen C, Rohrer C, Roth A, Gabriel H, Barz D, Gruen M. Vaccenic acid-mediated reduction in cytokine production is independent of c9,t11-CLA in human peripheral blood mononuclear cells. Biochim Biophys Acta. 2012 Oct;1821(10):1316-22. doi: 10.1016/j.bbalip.2012.06.010. Epub 2012 Jun 30. PMID 22750019
- [Background] Huebner SM, Olson JM, Campbell JP, Bishop JW, Crump PM, Cook ME. Low Dietary c9t11-Conjugated Linoleic Acid Intake from Dairy Fat or Supplements Reduces Inflammation in Collagen-Induced Arthritis. Lipids. 2016 Jul;51(7):807-19. doi: 10.1007/s11745-016-4163-8. Epub 2016 Jun 7. PMID 27270404
- [Background] Penedo LA, Nunes JC, Gama MA, Leite PE, Quirico-Santos TF, Torres AG. Intake of butter naturally enriched with cis9,trans11 conjugated linoleic acid reduces systemic inflammatory mediators in healthy young adults. J Nutr Biochem. 2013 Dec;24(12):2144-51. doi: 10.1016/j.jnutbio.2013.08.006. PMID 24231103
- [Background] Reynolds CM, Roche HM. Conjugated linoleic acid and inflammatory cell signalling. Prostaglandins Leukot Essent Fatty Acids. 2010 Apr-Jun;82(4-6):199-204. doi: 10.1016/j.plefa.2010.02.021. Epub 2010 Mar 7. PMID 20207526
- [Background] Stachowska E, Siennicka A, Baskiewcz-Halasa M, Bober J, Machalinski B, Chlubek D. Conjugated linoleic acid isomers may diminish human macrophages adhesion to endothelial surface. Int J Food Sci Nutr. 2012 Feb;63(1):30-5. doi: 10.3109/09637486.2011.593505. Epub 2011 Jul 1. PMID 21721848
- [Background] Viladomiu M, Hontecillas R, Bassaganya-Riera J. Modulation of inflammation and immunity by dietary conjugated linoleic acid. Eur J Pharmacol. 2016 Aug 15;785:87-95. doi: 10.1016/j.ejphar.2015.03.095. Epub 2015 May 15. PMID 25987426
- [Background] Poudel-Tandukar K, Nanri A, Matsushita Y, Sasaki S, Ohta M, Sato M, Mizoue T. Dietary intakes of alpha-linolenic and linoleic acids are inversely associated with serum C-reactive protein levels among Japanese men. Nutr Res. 2009 Jun;29(6):363-70. doi: 10.1016/j.nutres.2009.05.012. PMID 19628101
- [Background] Reifen R, Karlinsky A, Stark AH, Berkovich Z, Nyska A. alpha-Linolenic acid (ALA) is an anti-inflammatory agent in inflammatory bowel disease. J Nutr Biochem. 2015 Dec;26(12):1632-40. doi: 10.1016/j.jnutbio.2015.08.006. Epub 2015 Aug 14. PMID 26350254
- [Background] Ren J, Chung SH. Anti-inflammatory effect of alpha-linolenic acid and its mode of action through the inhibition of nitric oxide production and inducible nitric oxide synthase gene expression via NF-kappaB and mitogen-activated protein kinase pathways. J Agric Food Chem. 2007 Jun 27;55(13):5073-80. doi: 10.1021/jf0702693. Epub 2007 Jun 2. PMID 17542608
- [Background] Zhao G, Etherton TD, Martin KR, Gillies PJ, West SG, Kris-Etherton PM. Dietary alpha-linolenic acid inhibits proinflammatory cytokine production by peripheral blood mononuclear cells in hypercholesterolemic subjects. Am J Clin Nutr. 2007 Feb;85(2):385-91. doi: 10.1093/ajcn/85.2.385. PMID 17284733
- [Background] Mika A, Stepnowski P, Kaska L, Proczko M, Wisniewski P, Sledzinski M, Sledzinski T. A comprehensive study of serum odd- and branched-chain fatty acids in patients with excess weight. Obesity (Silver Spring). 2016 Aug;24(8):1669-76. doi: 10.1002/oby.21560. Epub 2016 Jun 29. PMID 27355152
- [Background] Rodriguez JM, Murphy K, Stanton C, Ross RP, Kober OI, Juge N, Avershina E, Rudi K, Narbad A, Jenmalm MC, Marchesi JR, Collado MC. The composition of the gut microbiota throughout life, with an emphasis on early life. Microb Ecol Health Dis. 2015 Feb 2;26:26050. doi: 10.3402/mehd.v26.26050. eCollection 2015. PMID 25651996
- [Background] Salminen S, Gibson GR, McCartney AL, Isolauri E. Influence of mode of delivery on gut microbiota composition in seven year old children. Gut. 2004 Sep;53(9):1388-9. doi: 10.1136/gut.2004.041640. No abstract available. PMID 15306608
- [Background] Moreno-Indias I, Cardona F, Tinahones FJ, Queipo-Ortuno MI. Impact of the gut microbiota on the development of obesity and type 2 diabetes mellitus. Front Microbiol. 2014 Apr 29;5:190. doi: 10.3389/fmicb.2014.00190. eCollection 2014. PMID 24808896
- [Background] Mai V, Draganov PV. Recent advances and remaining gaps in our knowledge of associations between gut microbiota and human health. World J Gastroenterol. 2009 Jan 7;15(1):81-5. doi: 10.3748/wjg.15.81. PMID 19115471
- [Background] Lozupone CA, Stombaugh JI, Gordon JI, Jansson JK, Knight R. Diversity, stability and resilience of the human gut microbiota. Nature. 2012 Sep 13;489(7415):220-30. doi: 10.1038/nature11550. PMID 22972295
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Festi D, Schiumerini R, Eusebi LH, Marasco G, Taddia M, Colecchia A. Gut microbiota and metabolic syndrome. World J Gastroenterol. 2014 Nov 21;20(43):16079-94. doi: 10.3748/wjg.v20.i43.16079. PMID 25473159
- [Background] Graf D, Di Cagno R, Fak F, Flint HJ, Nyman M, Saarela M, Watzl B. Contribution of diet to the composition of the human gut microbiota. Microb Ecol Health Dis. 2015 Feb 4;26:26164. doi: 10.3402/mehd.v26.26164. eCollection 2015. PMID 25656825
- [Background] Zimmer J, Lange B, Frick JS, Sauer H, Zimmermann K, Schwiertz A, Rusch K, Klosterhalfen S, Enck P. A vegan or vegetarian diet substantially alters the human colonic faecal microbiota. Eur J Clin Nutr. 2012 Jan;66(1):53-60. doi: 10.1038/ejcn.2011.141. Epub 2011 Aug 3. PMID 21811294
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Caesar R, Tremaroli V, Kovatcheva-Datchary P, Cani PD, Backhed F. Crosstalk between Gut Microbiota and Dietary Lipids Aggravates WAT Inflammation through TLR Signaling. Cell Metab. 2015 Oct 6;22(4):658-68. doi: 10.1016/j.cmet.2015.07.026. Epub 2015 Aug 27. PMID 26321659
- [Background] Caesar R, Nygren H, Oresic M, Backhed F. Interaction between dietary lipids and gut microbiota regulates hepatic cholesterol metabolism. J Lipid Res. 2016 Mar;57(3):474-81. doi: 10.1194/jlr.M065847. Epub 2016 Jan 18. PMID 26783361
- [Background] Walsh, H. H., H.; Cersosimo, L.; Kien, C.L.; Kraft, J. Decreased abundance of firmicutes in the gut microbiota after consumption of a diet containing milk fats. FASEB J 30, 683.611 (2016).
- [Derived] Taormina VM, Eisenhardt S, Gilbert MP, Poynter ME, Kien CL, Kraft J. Full-fat yogurt compared with non-fat yogurt reduces blood triacylglycerol concentrations and lowers the triacylglycerol content in specific lipoprotein subclasses in adults with prediabetes: an exploratory analysis of a randomized-controlled trial. Lipids Health Dis. 2025 Jun 5;24(1):201. doi: 10.1186/s12944-025-02616-4. PMID 40474187
- [Derived] Taormina VM, Eisenhardt S, Gilbert MP, Poynter ME, Kien CL, Kraft J. Full-fat versus non-fat yogurt consumption improves glucose homeostasis and metabolic hormone regulation in individuals with prediabetes: A randomized-controlled trial. Nutr Res. 2025 Apr;136:39-52. doi: 10.1016/j.nutres.2025.02.005. Epub 2025 Feb 28. PMID 40139076